CLINICAL TRIAL: NCT07099274
Title: A Single-Arm, Single-Center Clinical Study Evaluating the Efficacy and Safety of Lparomlimab and Tuvonralimab Injection in Combination With TACE and Lenvatinib as Second-Line Therapy for Unresectable Intermediate-to-Advanced Hepatocellular Carcinoma
Brief Title: Lparomlimab and Tuvonralimab Injection in Combination With TACE and Lenvatinib in the Treatment of Second-Line Therapy for Unresectable Intermediate-to-Advanced Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC-2025-0041
Record Dates: First submitted 2025-07-13; First posted 2025-08-01 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-07

CONDITIONS: HCC
Keywords: Iparomlimab and Tuvonralimab Injection; TACE; Lenvatinib
MeSH Terms: interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- lparomlimab and Tuvonralimab Injection in Combination with TACE and Lenvatinib (Experimental): lparomlimab and Tuvonralimab Injection in Combination with TACE and Lenvatinib
  Interventions: Drug: lparomlimab and Tuvonralimab Injection in Combination with TACE and Lenvatinib

INTERVENTIONS:
Drug: lparomlimab and Tuvonralimab Injection in Combination with TACE and Lenvatinib — lparomlimab and Tuvonralimab Injection (QL1706): 7.5 mg/kg, q3w; Lenvatinib: 8 mg once daily for patients weighing <60 kg, or 12 mg once daily for those weighing ≥60 kg, administered orally, continuous daily dosing； TACE: Administered 4-6 times, using a combination of anthracyclines, lipiodol, and microspheres. The procedure should be performed within one week before or after QL1706 administration.

SUMMARY:
Major objectives To evaluate the efficacy of lparomlimab and Tuvonralimab injection (QL1706, an Anti-PD-1/ CTLA-4 Combined Antibody) in combination with TACE and lenvatinib as second-line therapy in patients with unresectable intermediate-to-advanced hepatocellular carcinoma.

DETAILED DESCRIPTION:
This single-arm, single-center clinical study aims to evaluate the efficacy and safety of lparomlimab and Tuvonralimab injection (QL1706, an Anti-PD-1/ CTLA-4 Combined Antibody) in combination with TACE and lenvatinib as second-line therapy in patients with unresectable intermediate-to-advanced hepatocellular carcinoma. This study consists of three phases: screening, treatment, and follow-up. Efficacy evaluation and safety monitoring should be performed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Comprehension and voluntary signing of the study's informed consent form;
* Age ≥18 years, any gender;
* Histologically or clinically confirmed hepatocellular carcinoma;
* Documented failure or intolerance to first-line therapy with PD-1/PD-L1 inhibitor plus bevacizumab;
* ECOG performance status 0-2;
* Child-Pugh class A or class B (score ≤7) without hepatic encephalopathy history;
* Life expectancy ≥3 months;
* At least one measurable target lesion confirmed by screening imaging per RECIST v1.1;
* Adequate organ and bone marrow function within 7 days prior to initial study treatment;
* Active HBV/HCV infection requires ongoing antiviral therapy; k.Fertile patients must use highly effective contraception with partners during treatment and ≥180 days post-last dose.

  2.Exclusion Criteria:
* Inability to comply with the study protocol or procedures;
* Histologically/cytologically confirmed fibrolamellar HCC, sarcomatoid HCC, cholangiocarcinoma, or mixed hepatocellular-cholangiocarcinoma;
* History of liver transplantation or planned transplantation;
* Presence of central nervous system metastases and/or leptomeningeal carcinomatosis;
* Baseline imaging showing Vp4 portal vein tumor thrombosis;
* Hypersensitivity to any study drug components or history of severe allergic reactions;
* Concurrent HBV and HCV co-infection;
* Clinically significant ascites requiring intervention during screening;
* Concurrent use of other investigational drugs or participation in another clinical trial within 4 weeks prior to enrollment;
* Esophageal/gastric variceal bleeding due to portal hypertension within 6 months before treatment initiation, or high-risk varices on endoscopy within 3 months;
* Current interstitial lung disease (ILD), history of steroid-required ILD, or other pulmonary fibrosis/organizing pneumonia affecting immune-related pulmonary toxicity assessment;
* Uncontrolled hypertension (SBP≥160 mmHg and/or DBP≥100 mmHg despite medication), coronary artery disease, arrhythmias, or heart failure (NYHA Class ≥II);
* Uncontrolled clinically significant infections requiring IV antimicrobial therapy;
* Proteinuria ≥2+ (≥1.0g/24h);
* History of hemorrhagic tendency regardless of severity within 2 months prior to enrollment;
* Arterial/venous thromboembolic events within 12 months before treatment initiation (e.g., cerebrovascular accident including TIA);
* Acute myocardial infarction, acute coronary syndrome, or CABG within 6 months before treatment;
* Unhealed fractures or chronic non-healing wounds;
* Coagulopathy, bleeding diathesis, or current therapeutic anticoagulation;
* Other malignancies within 5 years except curatively resected basal/squamous cell skin carcinoma or cervical carcinoma in situ;
* Active autoimmune disease or autoimmune disease history requiring immunosuppression within 4 weeks prior to enrollment;
* Prior allogeneic bone marrow or solid organ transplantation;
* Investigator assessment of ineligibility based on medical/safety reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2025-08-22 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | up to 12 month
  PFS was defined as the time from first dose of study treatment to the first documented PD per RECIST 1.1 by investigator assessment, or death due to any cause, whichever occurred first.

SECONDARY OUTCOMES:
Objective response rate | up to 12 month
  the percentage of participants in the analysis population who had a CR (Disappearance of all target lesions) or a PR (≥30% decrease in SOD of target lesions) using RECIST 1.1 based on investigator assessment.
Overall survival | up to 36 month
  OS was defined as the time from the first dose of study drug to death due to any cause.
Disease Control Rate | up to 12 month
  DCR was defined as the percentage of participants in the analysis population who have CR (Disappearance of all target lesions) or PR (≥30% decrease in SOD of target lesions) or SD (Neither sufficient shrinkage for PR nor sufficient increase for PD [at ≥20% increase in target lesion SOD and absolute SOD increase of ≥5 mm.
Duration of Response | up to 12 month
  For participants who demonstrated a confirmed CR (disappearance of all target lesions) or PR (≥30% decrease in SOD of target lesions) per RECIST 1.1 by investigator assessment, DOR was defined as time from first documented CR or PR until PD or death, whichever occurs first.
Adverse Events | up to 36 month
  An AE was defined as any untoward medical occurrence in a pharmaceutical product which does not necessarily have to have a causal relationship with this treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No